CLINICAL TRIAL: NCT01629329
Title: A Randomized, Double-blind Comparison of Single Dose Prochlorperazine Versus Acetaminophen, Aspirin and Caffeine for the Treatment of Acute Migraine in the Emergency Department.
Brief Title: Prochlorperazine Versus Acetaminophen, Aspirin, and Caffeine for the Treatment of Acute Migraine
Acronym: Migraine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no difference found between two groups in a preliminary analysis
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4258
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2014-06

CONDITIONS: Migraine Headaches
Keywords: Headache; prochlorperazine; excedrin migraine; treatment efficacy; pain scores
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Aspirin; Acetaminophen; acetaminophen, aspirin, caffeine drug combination; Prochlorperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin, Acetaminophen, Caffeine pills (Active Comparator): Patients receiving AAC(acetaminophen 250mg, aspirin 250mg and caffeine 65mg in each tablet)will receive 2 pills with active compound and placebo syringe with 2 ml of saline.
  Interventions: Drug: Aspirin, Acetaminophen, Caffeine pills
- Prochlorperazine 10mg (Active Comparator): Patients will receive active compound of Prochlorperazine 10mg via IV syringe and 2 unmarked placebo pills
  Interventions: Drug: Prochlorperazine 10mg

INTERVENTIONS:
Drug: Aspirin, Acetaminophen, Caffeine pills — One time dose of 2 pills each containing acetaminophen 250mg, aspirin 250mg and caffeine 65mg in each tablet. Simultaneous administration of placebo(5ml of saline administered IV)
  Other Names: Excedrin
  Arms: Aspirin, Acetaminophen, Caffeine pills
Drug: Prochlorperazine 10mg — One time dose of Prochlorperazine 10mg/2ml given IV slow push. Simultaneous administration of 2 unmarked placebo pills.
  Other Names: Compazine
  Arms: Prochlorperazine 10mg

SUMMARY:
The objective of this randomized, double blind study is to demonstrate that one dose oral "excedrin migraine" (acetaminophen, aspirin and caffeine) is not inferior when compared to one dose of intravenous prochlorperazine for the treatment of acute migraine headaches in the emergency department.

DETAILED DESCRIPTION:
Patients with severe headaches often come to the emergency department seeking relief from their symptoms. There is some dating suggesting that over the counter treatment options are not inferior to treatment options offered in emergency departments. Patients presenting to the Einstein Emergency Department with IHS criteria for migraine headache will be approached by research associate and offered to participate in a randomized double blind study comparing excedrin migraine to compazine. Patients will be randomized by the hospital pharmacy. The pharmacy will distribute one of two packets, one containing prochlorperazine 10mg and 2 placebo tablets, the other containing 2 generic AAC tablets without scoring (acetaminophen 250mg, aspirin 250mg and caffeine 65mg in each tablet) and a placebo syringe. Patients will be monitored for improvement of pain, change in vital signs, and adverse events for two hours after receiving drugs. At 24 hours, the patients will be called back to access if they experienced any side effects from the time of discharge, and if they would take this medicine again if they experienced another migraine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Headache must meet the IHS criteria for migraine or probable migraine

  * 2 out of 4 of following:

    * Unilateral location
    * Throbbing (pulsating) quality
    * Moderate to severe intensity (inhibits/prohibits daily activities)
    * Exacerbation with moderate activity or mild activity
  * During HA, at least 1 out of 3 of following:

    * Nausea and/or vomiting
    * Photophobia
    * Phonophobia

Exclusion Criteria:

* Known allergy to study medications
* Pregnancy
* < 18 years old
* Inability to provide written, informed consent
* Patients with positive lumbar puncture or positive CT scan for suspected secondary headache
* History of peptic ulcer disease
* History of liver failure
* History of coagulopathy
* Gastrointestinal bleeding within the last 3 months
* Previous gastrointestinal bleeding with non-steroidal anti-inflammatory medications
* Ingestion of other pain medications within the previous six hours deemed to put the patient at risk of exceeding a toxic dose of ASA or acetaminophen (> 100mg/kg for ASA or acetaminophen)
* Vomiting within one hour of receiving oral study medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-11; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Deitch, DO, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Pre-assignment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Period: Overall Study
Arm/Group | Aspirin, Acetaminophen, Caffeine Pills | Prochlorperazine 10mg
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin, Acetaminophen, Caffeine Pills | Prochlorperazine 10mg | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference From Baseline of VAS Pain Scores
Description: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Time Frame: 60 minutes from drug administration
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Aspirin, Acetaminophen, Caffeine Pills | Prochlorperazine 10mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Reported Adverse Side-effects
Description: Secondary endpoints will also be assessed at 30min, 90min and 120min. Additional secondary endpoints will be in the number of reported adverse side-effects, defined as muscle spasm, tiredness, extreme restlessness, GI upset, vomiting in the ED and treatment failure rate.
Time Frame: 30, 90, and 120 minutes from drug administration
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Aspirin, Acetaminophen, Caffeine Pills | Prochlorperazine 10mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Description: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Aspirin, Acetaminophen, Caffeine Pills | Prochlorperazine 10mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes